CLINICAL TRIAL: NCT06366451
Title: A Phase 0 Multicenter Study of the Pharmacodynamic Effects of Intratumoral Microdose Administration of Rilvegostomig, Volrustomig, Sabestomig, and AZD9592
Brief Title: PBI-MST-01 (NCT04541108) Substudy AZN-05: Intratumoral Microdosing of Rilvegostomig, Volrustomig, Sabestomig, and AZD9592 in HNSCC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Presage Biosciences (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MST01-AZN-05; PBI-MST-01 (Other: Presage Biosciences)
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; intratumoral microdosing; microdose injection; microdosing; in vivo oncology; tumor microenvironment; multiplexed immunohistochemistry; head and neck cancer; head and neck squamous cell carcinoma; pharmacodynamic biomarkers; CIVO; master protocol; precision oncology; spatial biology
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is an exploratory clinical trial to evaluate intratumoral mechanistic effects of novel and approved agents on intact human tumors. This is a cohort substudy of a Master Protocol (PBI-MST-01, NCT04541108) framework, under which comparisons will not be made between substudy cohorts.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rilvegostomig, Volrustomig, Sabestomig, AZD9592, Pembrolizumab (Experimental): HNSCC patients presenting with a surface accessible lesion who are scheduled for tumor and/or regional node dissection as part of their standard treatment will be injected one to three days prior to surgery using the CIVO device. The planned injection scheme includes: vehicle control and microdoses of rilvegostomig, volrustomig, sabestomig, AZD9592, and pembrolizumab as single agents and AZD9592 drug combinations with the evaluated biologics.
  Interventions: Biological: Rilvegostomig; Biological: Volrustomig; Biological: Sabestomig; Biological: AZD9592; Biological: Pembrolizumab; Combination Product: AZD9592 + Rilvegostomig; Combination Product: AZD9592 + Volrustomig; Combination Product: AZD9592 + Sabestomig; Combination Product: AZD9592 + Pembrolizumab

INTERVENTIONS:
Biological: Rilvegostomig — Intratumoral microdose injection by the CIVO device.
  Other Names: AZD2936
Biological: Volrustomig — Intratumoral microdose injection by the CIVO device.
  Other Names: MEDI5752
Biological: Sabestomig — Intratumoral microdose injection by the CIVO device.
  Other Names: AZD7789
Biological: AZD9592 — Intratumoral microdose injection by the CIVO device.
Biological: Pembrolizumab — Intratumoral microdose injection by the CIVO device.
  Other Names: Keytruda, MK-3475
Combination Product: AZD9592 + Rilvegostomig — Intratumoral microdose injection by the CIVO device.
Combination Product: AZD9592 + Volrustomig — Intratumoral microdose injection by the CIVO device.
Combination Product: AZD9592 + Sabestomig — Intratumoral microdose injection by the CIVO device.
Combination Product: AZD9592 + Pembrolizumab — Intratumoral microdose injection by the CIVO device.

SUMMARY:
This is a multi-center, open-label, Phase 0 substudy designed to evaluate the localized pharmacodynamics (PD) of rilvegostomig, volrustomig, sabestomig, and AZD9592 within the tumor microenvironment (TME) when administered intratumorally in microdose quantities via the CIVO device in patients presenting with Head and Neck Squamous Cell Carcinoma (HNSCC) with a surface accessible lesion, who are scheduled for tumor and/or regional node dissection as part of their standard treatment. PD effects due to injected investigational agents, either as single agents or as AZD9592 drug combinations with the evaluated biologics, will be compared to those elicited by pembrolizumab alone, which will also be injected in microdose quantities via the CIVO device.

DETAILED DESCRIPTION:
The CIVO Microdose Injection Device (MID) simultaneously delivers multiple drugs and drug combinations (Up to 8), each in microdose amounts, into a single patient tumor and enables comparisons of the resulting biomarker responses that occurred while that tumor was still in the native microenvironment. AstraZeneca is developing three novel assets: rilvegostomig, volrustomig, and sabestomig, all of which are bispecific monoclonal antibodies designed to stimulate antitumor immunity. In this Phase 0 clinical trial, the PD effects of these investigational assets in the TME of patients presenting with HNSCC will be evaluated. These investigational assets will be injected alone in microdose quantities at tumor sites in HNSCC patients. Pembrolizumab, also used therapeutically in this patient population, will be included in the CIVO injection array administered as a single agent. In addition, microdoses of AZD9592, a novel antibody drug conjugate (ADC), alone or in combinations with the evaluated biologics will also be assessed. The CIVO-injected portion of the tissue will be analyzed for localized response at sites of drug exposure in the TME.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide written informed consent. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
2. Male or female ≥ 18 years of age at Visit 1 (Screening).
3. Pathologic diagnosis of Head and Neck Squamous Cell Carcinoma (HNSCC) of the oropharynx, hypopharynx, oral cavity, or larynx.
4. Ability and willingness to comply with the study's visits and assessment schedule.
5. At least one lesion (primary tumor, recurrent tumor, metastasis, or metastatic lymph node) that is surface accessible for CIVO injection that contains viable minimum tumor tissue volume and characteristics (e.g., based on clinical evaluation, available pre-operative imaging, pre-injection ultrasound imaging, or pathology reports indicating lesion with appropriate viable tumor volume without excessive cysts or necrosis) and for which there is a planned surgical intervention. The patient's presentation, surgical and pathology plan may determine whether a lesion is eligible with respect to a given CIVO MID needle configuration.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Female patients who:

   * Are postmenopausal for at least one year before the screening visit, OR
   * Are surgically sterile, OR
   * Are of childbearing potential who agree to practice a highly effective method of contraception from the time of signing the Informed Consent Form (ICF) until 7 months after the CIVO injection OR agree to completely abstain from heterosexual intercourse.
   * Agree to refrain from donating, or retrieving for their own use, ova until 7 months after the CIVO injection.
   * Agree to refrain from breastfeeding until 7 months after the CIVO injection.
8. Male patients, even if surgically sterile (i.e., status post-vasectomy), who:

   * Agree to practice effective barrier contraception from the time of signing the ICF until 7 months after the CIVO injection OR agree to completely abstain from heterosexual intercourse.
   * Agree to refrain from fathering a child or donating sperm until 7 months after the CIVO injection.

Exclusion Criteria:

1. Tumors and/or effaced nodes that are anticipated by the Investigator to lack a sufficient volume of viable tumor tissue (Based on available pre-operative imaging, pre-injection ultrasound imaging, or pathology reports) for CIVO microdose injection due to necrosis, cysts, excessive stroma, fibrosis, or treatment-induced tissue changes.
2. Tumors near or involving critical structures for which, in the opinion of the treating clinician, injection would pose undue risk to the patient.
3. Prior exposure to immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies within the last 5 years.
4. Previous treatment with another ADC containing a chemotherapeutic agent that inhibits topoisomerase 1 activity or with another epidermal growth factor receptor (EGFR) and/or mesenchymal-epithelial transition factor (c-MET) targeted ADC.
5. Patients with concurrent cancer, immune disease or active infection requiring systemic or radiotherapy.
6. Female patients who:

   * Intend to become pregnant during the study,
   * Are both lactating and breastfeeding, OR
   * Have a positive beta-subunit human chorionic gonadotropin (beta-hCG) pregnancy test at screening verified by the Investigator.
7. Any uncontrolled intercurrent illness, condition, serious medical or psychiatric illness, or circumstance that, in the opinion of the Investigator, could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives.
8. History of organ transplant.
9. Major surgery within 4 weeks prior to injection: subject must have adequate wound healing and have recovered from any prior surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of signature scores using Gene Set Variability Analysis within regions injected with microdoses of rilvegostomig, volrustomig, sabestomig, AZD9592, or pembrolizumab as single agents or as AZD9592 drug combinations with the evaluated biologics | 1 to 3 days after microdose injection
  The localized activity of injected microdoses will be analyzed using the NanoString GeoMx Digital Spatial Profiler (DSP) and the GeoMx Cancer Transcriptome Atlas to comprehensively profile over 1800 genes simultaneously with spatial resolution to describe tumor biology, the TME, and the immune response signatures of each drug at an injection site. DSP outcomes may be validated via IHC, immunofluorescence, or ISH technique.

SECONDARY OUTCOMES:
Incidence of reported Adverse Events and/or Adverse Device Effects [Safety and Tolerability] | Up to 28 days after microdose injection
  Safety of the microdose injection procedure and injected content will be assessed by quantification of the frequency, intensity, and relatedness of all reported Adverse Events and/or Adverse Device Effects.

OTHER OUTCOMES:
Evaluation of tumor whole exome sequencing (WES)/whole transcriptome sequencing (WTS) | Sample collected at screening
  Tumor WES/WTS will be performed to help develop a comprehensive understanding of the observed PD responses of the tumor samples to the injected microdoses of the study drugs. Tumor WES/WTS (with matched blood circulating tumor DNA as control) will collect information on the tumor and TME background to provide critical tumor- and immune-related information such as, but not limited to, T-cell and B-cell repertoire, microsatellite instability, tumor mutational burden, and immunogenomic changes/immune profiling of the TME.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Presage Biosciences
Locations (7):
- United States (7):
  - UC Davis, Sacramento, California
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derry JMJ, Burns C, Frazier JP, Beirne E, Grenley M, DuFort CC, Killingbeck E, Leon M, Williams C, Gregory M, Houlton J, Clayburgh D, Swiecicki P, Huszar D, Berger A, Klinghoffer RA. Trackable Intratumor Microdosing and Spatial Profiling Provide Early Insights into Activity of Investigational Agents in the Intact Tumor Microenvironment. Clin Cancer Res. 2023 Sep 15;29(18):3813-3825. doi: 10.1158/1078-0432.CCR-23-0827. PMID 37389981
- [Background] Gundle KR, Deutsch GB, Goodman HJ, Pollack SM, Thompson MJ, Davis JL, Lee MY, Ramirez DC, Kerwin W, Bertout JA, Grenley MO, Sottero KHW, Beirne E, Frazier J, Dey J, Ellison M, Klinghoffer RA, Maki RG. Multiplexed Evaluation of Microdosed Antineoplastic Agents In Situ in the Tumor Microenvironment of Patients with Soft Tissue Sarcoma. Clin Cancer Res. 2020 Aug 1;26(15):3958-3968. doi: 10.1158/1078-0432.CCR-20-0614. Epub 2020 Apr 16. PMID 32299817
- [Background] Klinghoffer RA, Bahrami SB, Hatton BA, Frazier JP, Moreno-Gonzalez A, Strand AD, Kerwin WS, Casalini JR, Thirstrup DJ, You S, Morris SM, Watts KL, Veiseh M, Grenley MO, Tretyak I, Dey J, Carleton M, Beirne E, Pedro KD, Ditzler SH, Girard EJ, Deckwerth TL, Bertout JA, Meleo KA, Filvaroff EH, Chopra R, Press OW, Olson JM. A technology platform to assess multiple cancer agents simultaneously within a patient's tumor. Sci Transl Med. 2015 Apr 22;7(284):284ra58. doi: 10.1126/scitranslmed.aaa7489. PMID 25904742
- [Background] Frazier JP, Bertout JA, Kerwin WS, Moreno-Gonzalez A, Casalini JR, Grenley MO, Beirne E, Watts KL, Keener A, Thirstrup DJ, Tretyak I, Ditzler SH, Tripp CD, Choy K, Gillings S, Breit MN, Meleo KA, Rizzo V, Herrera CL, Perry JA, Amaravadi RK, Olson JM, Klinghoffer RA. Multidrug Analyses in Patients Distinguish Efficacious Cancer Agents Based on Both Tumor Cell Killing and Immunomodulation. Cancer Res. 2017 Jun 1;77(11):2869-2880. doi: 10.1158/0008-5472.CAN-17-0084. Epub 2017 Mar 31. PMID 28364003
- [Background] Dey J, Kerwin WS, Grenley MO, Casalini JR, Tretyak I, Ditzler SH, Thirstrup DJ, Frazier JP, Pierce DW, Carleton M, Klinghoffer RA. A Platform for Rapid, Quantitative Assessment of Multiple Drug Combinations Simultaneously in Solid Tumors In Vivo. PLoS One. 2016 Jun 30;11(6):e0158617. doi: 10.1371/journal.pone.0158617. eCollection 2016. PMID 27359113
- [Background] Moreno-Gonzalez A, Olson JM, Klinghoffer RA. Predicting responses to chemotherapy in the context that matters - the patient. Mol Cell Oncol. 2015 Jun 10;3(1):e1057315. doi: 10.1080/23723556.2015.1057315. eCollection 2016 Jan. PMID 27308571